CLINICAL TRIAL: NCT00125294
Title: Evaluation of a Dose Titration Protocol for Sublingual Methadone Hydrochloride for the Management of Cancer-related Breakthrough Pain
Brief Title: Sublingual Methadone for the Management of Cancer Breakthrough Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Calgary Health Region (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17208; Calgary Health Region
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2011-08

CONDITIONS: Cancer; Pain
Keywords: cancer pain; breakthrough pain; methadone; dose titration; sublingual route of administration; Cancer related pain; currently taking narcotics
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain; Breakthrough Pain | interventions — Methadone

INTERVENTIONS:
Drug: Methadone

SUMMARY:
A dose titration protocol for sublingual methadone hydrochloride for the management of cancer-related breakthrough pain to find the optimal dose.

DETAILED DESCRIPTION:
This is a dose titration protocol for sublingual methadone hydrochloride for the management of cancer-related breakthrough pain to find the optimal dose.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Experiences episodes of breakthrough pain which respond to opioid therapy
* Controlled baseline pain
* Cognitive status sufficient for accurate completion of assessment form
* Willing to provide written informed consent
* Ability to hold a volume of 1 cc of water under the tongue for 5 minutes

Exclusion Criteria:

* Currently or has received methadone during the previous week
* Recent history of substance abuse
* Severe respiratory impairment or other contraindications to opioids
* Recently received therapies that had the potential to alter pain intensity or response to analgesics
* Symptomatic anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-09; Primary Completion 2006-06 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Determine optimal dose titration
Determine assessment protocol

CONTACTS AND LOCATIONS:
Overall Officials: Neil Hagen, Principal Investigator — Alberta Cancerboard